CLINICAL TRIAL: NCT02321371
Title: Effect of Goal Directed Ammonia Lowering Therapy in Acute on Chronic Liver Failure Patients With Hepatic Encephalopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-HE-01
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2017-01

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Lactulose; Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lactulose + Rifaximin (Experimental): Continuation of Lactulose + addition of Rifaximin 400 mg 8th hourly through enteral route.
  Interventions: Drug: Lactulose + Rifaximin
- Lactulose therapy (Active Comparator)
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: Lactulose + Rifaximin — Lactulose + addition of Rifaximin 400 mg 8th hourly through enteral route
  Arms: Lactulose + Rifaximin
Drug: Lactulose — Continuation of Lactulose therapy for further 48 hours.
  Arms: Lactulose therapy

SUMMARY:
In this study, all patients with ACLF (Acute on Chronic Liver Failure) with grade III/IV HE (Hepatic Encephalopathy) getting admitted in our institute will be enrolled after the fulfilment of inclusion/exclusion criteria and consent of the patient's attendants. Investigation of the patient (as mentioned in the proforma) will be done.

Intervention step 1:

liq Lactulose 100 mL stat followed by 30 mL/ hourly through NG/NJ route + Lactulose enema 3rd hourly - till 4 time soft stool is passed, then 30 mL through enteral route 6th hourly (If patient has no bowel sounds, only enema will be given)

Intervention step 2:

(after 24 hours of introduction of step 1, if no rapid reduction in ammonia to <70mcg/dL) Randomization to L or R arm R Arm (Addition of Rifaximin) Continuation of Lactulose + addition of Rifaximin 400 mg 8th hourly through enteral route L Arm (Lactulose only) Continuation of Lactulose therapy for further 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Patients with ACLF with grade III/IV HE

Exclusion Criteria:

1. Patients with prior decompensation
2. Grade I,II HE
3. Chronic HE
4. CV stroke
5. Patients with ammonia level <70 mcg/dL
6. Patients with Septic shock
7. Pregnant lady

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-10-19 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Reduction of ammonia level to <70 mcg/dL within 72 hours of the ammonia reduction treatment. | 3 days

SECONDARY OUTCOMES:
Reduction of ammonia level to at least 50% of the baseline value within 72 hours. | 3 days
Duration of hepatic encephalopathy post-inclusion. | 10 days
  10 days after enrollment or 7 days after achieving primary endpoint, whichever is shorter.
Improvement in hepatic encephalopathy from grade III-IV to II-I at any time within 72 hours of treatment. | 3 days
Liver disease related and overall mortality. | 10 days
  10 days after enrollment or 7 days after achieving primary endpoint, whichever is shorter.
Duration of ICU stay. | 10 days
  10 days after enrollment or 7 days after achieving primary endpoint, whichever is shorter.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tanmay Vyas, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Zacharias HD, Kamel F, Tan J, Kimer N, Gluud LL, Morgan MY. Rifaximin for prevention and treatment of hepatic encephalopathy in people with cirrhosis. Cochrane Database Syst Rev. 2023 Jul 19;7(7):CD011585. doi: 10.1002/14651858.CD011585.pub2. PMID 37467180